CLINICAL TRIAL: NCT00466661
Title: A Double-Blind, Randomized, Placebo-Controlled Trial of Acamprosate in Alcohol-Dependent Individuals With Comorbid Bipolar Disorder
Brief Title: Acamprosate vs. Placebo in Bipolar Alcoholics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR#16928
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Alcohol Dependence; Bipolar Disorder
Keywords: Acamprosate; Alcoholism; Bipolar disorder; Comorbidity; Craving; Depression; GABA; Glutamate; Mania; Pharmacotherapy; Withdrawal
MeSH Terms: conditions — Alcoholism; Bipolar Disorder; Depression; Mania | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acamprosate (Experimental): 666 mg p.o. TID
  Interventions: Drug: Acamprosate
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acamprosate — 666 mg po TID
  Arms: Acamprosate
Drug: Placebo — 2 tabs po TID
  Arms: Placebo

SUMMARY:
To conduct a double-blind, randomized, placebo-controlled outpatient clinical trial of acamprosate in individuals with alcohol dependence and bipolar disorder who are also receiving mood stabilizing medication. The study will assess the safety and efficacy of acamprosate in alcohol-dependent bipolar patients as measured by its effects on alcohol use and mood symptoms relative to placebo.

The primary hypothesis to be tested is whether individuals with comorbid bipolar disorder and alcohol dependence who receive acamprosate plus mood stabilizer will have greater improvement in alcohol-related outcomes than those who receive mood stabilizer alone. A secondary hypothesis that will be explored is that alcohol-dependent bipolar individuals treated with acamprosate will have greater mood stability as compared to those treated with mood stabilizers alone.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18-65
2. Meet DSM-IV criteria for current (past 90 days) alcohol dependence
3. Meet DSM-IV criteria for bipolar I or bipolar II disorder
4. Currently on a mood stabilizing medication regimen, including the use of lithium, valproic acid, lamotrigine, carbamazepine, and/or antipsychotic agent FDA approved to treat bipolar disorder without any dosage adjustments in the past 30 days
5. Must be able to remain free from alcohol for at least 3 days prior to medication initiation
6. Subjects must be able to adequately provide informed consent and function at an intellectual level sufficient to allow the accurate completion of all assessment instruments
7. Subjects must consent to random assignment and be willing to commit to medication treatment and follow-up assessments

Exclusion Criteria:

1. Individuals with a primary psychiatric disorder other than bipolar disorder
2. Individuals with an uncontrolled neurologic condition that could confound the results of the study
3. Individuals with an uncontrolled medical condition that may adversely affect the conduct of this trial or jeopardize the subject's safety
4. Participants with creatinine clearance less than or equal to half of normal value as indicated by chem. 7 results conducted at screening visit.
5. Concomitant use of other psychotropic medications not allowed per the protocol
6. Women of childbearing potential who are pregnant, lactating or refuse to use adequate forms of birth control
7. Current suicidal or homicidal risk
8. Baseline scores of > 35 on the Montgomery Asberg Depression Rating Scale and/or > 25 on the Young Mania Rating Scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan K Tolliver, M.D., Ph.D., Principal Investigator — Division of Clinical Neuroscience, Department of Psychiatry, Medical University of South Carolina; Kathleen T Brady, M.D., Ph.D., Study Director — Division of Clinical Neuroscience, Department of Psychiatry, Medical University of South Carolina
Locations (1):
- Institute of Psychiatry, Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment by clinical referral
Pre-assignment Details: Two week lead-in (Screening, Baseline)
Period: Overall Study
Arm/Group | Acamprosate | Placebo
Started | 16 | 17
At Least 1 Postrandomization Visit (Defines modified Intention to Treat (mITT) sample) | 14 | 16
Completed | 12 | 11
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acamprosate | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (6.7) | 43.7 (11.3) | 42.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Time to First Drink (Days)
Description: Number of days after randomization until consumption of first alcoholic beverage per self-report.
Time Frame: 8 weeks
Population: Sample analyzed is a modified intention to treat (mITT) sample of all randomized subjects who returned for at least one visit post-randomization (total mITT n=30).
Measure: Mean (95% Confidence Interval); unit: Days
Groups:
- Acamprosate: Participants assigned to acamprosate with at least one return visit after randomization
- Placebo: Participants assigned to placebo who returned for at least one visit after randomization
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 14 | 16
Days | 16.5 [6 to NA] — The upper range of the confidence interval was calculated to be infinity | 8.0 [2.0 to NA] — The upper range of the confidence interval was calculated to be infinity

2. Secondary Outcome: Percent Days Abstinent
Description: Percentage of days in trial with no alcohol consumption
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days in trial
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 14 | 16
percentage of days in trial | 77.0 (28.2) | 73.0 (29.5)

3. Secondary Outcome: Percent Heavy Drinking Days
Description: Percentage of drinking days that are heavy drinking days (5 or more standard drinks/day for males, 4 or more standard drinks/day for females)
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days drinking
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 14 | 16
percentage of days drinking | 6.4 (8.4) | 10.7 (14.6)

4. Secondary Outcome: Percent Carbohydrate-deficient Transferrin
Description: Measured level of validated serum alcohol biomarker
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: "percent CDT"
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 14 | 16
"percent CDT" | 2.4 (0.8) | 2.5 (1.8)

5. Secondary Outcome: Gamma-glutamyltransferase
Description: Measured levels of validated serum alcohol biomarker
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gamma-glutamyltransferase U/L
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 14 | 16
Gamma-glutamyltransferase U/L | 37.1 (40.0) | 63.8 (67.0)

6. Secondary Outcome: Obsessive Compulsive Drinking Scale Score
Description: Higher scores indicate worse outcome; minimum score = 0, maximum score = 40
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 14 | 16
score on a scale | 10.8 (9.5) | 15.3 (12.3)

7. Secondary Outcome: Montgomery Asberg Depression Rating Scale Score
Description: MADRS scores at study endpoint. Higher scores indicate a worse outcome. Minimum score = 0, maximum score = 60.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 14 | 16
score on a scale | 8.7 (6.5) | 11.3 (8.5)

8. Secondary Outcome: Young Mania Rating Scale Score
Description: YMRS scores at study endpoint. Higher scores indicate a worse outcome. Minimum score = 0, maximum score = 60.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 14 | 16
score on a scale | 5.3 (2.9) | 5.4 (3.4)

9. Secondary Outcome: Clinical Global Impression Scale Score
Description: Higher values indicate worse outcomes; minimum value = 1, maximum value = 7
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acamprosate | Placebo
Number analyzed (Participants) | 14 | 16
score on a scale | 2.7 (1.4) | 3.7 (1.1)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Known adverse events and or serious adverse events are reported for a modified intention to treat (mITT) sample of all randomized subjects who returned for at least one visit post-randomization (total mITT n=30). Adverse event data (all-cause mortality, serious adverse events, all other adverse events) could not be obtained in randomized participants lost to follow-up (n=3).
Groups:
- Acamprosate: Participants assigned to acamprosate
- Placebo: Participants assigned to placebo
Arm/Group | Acamprosate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 3/14 | 3/16
Other Adverse Events (participants affected / at risk) | 6/14 | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acamprosate (N=14) | Placebo (N=16)
Hospitalization (Psychiatric disorders) | 2 (2) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Anaphylactoid skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acamprosate (N=14) | Placebo (N=16)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Headache (General disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diffuse aches (General disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Limited sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No